CLINICAL TRIAL: NCT03549325
Title: A Human Controlled Infection Study to Assess Colonisation and Immunogenicity Following Nasal Inoculation With Neisseria Lactamica With Eradication on Day 4 or 14
Brief Title: A Study Assessing Colonisation & Immunogenicity After Nasal Inoculation With N. Lactamica and Eradication on Day 4 or 14
Acronym: Lac-3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was paused in March 2020 due to the COVID pandemic. An interim data analysis was conducted in 2021 which confirmed that sufficient data had been collected to meet the primary objective, therefore the study was terminated.
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MED1354
Record Dates: First submitted 2017-10-23; First posted 2018-06-08 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Meningitis, Meningococcal
Keywords: Neisseria lactamica; healthy volunteers; nasal inoculation; colonisation
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Intervention Model Description: Group 1: Nasal inoculation with Neisseria lactamica with eradication on day 4 - up to 22 volunteers or until 11 colonised on day 4 Group 2: Nasal inoculation with Neisseria lactamica with eradication on day 14 - up to 22 volunteers or until 11 colonised on day 4
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Nasal drops containing Neisseria lactamica are administered at Day 0 by the study doctor.
  Eradication therapy with the antibiotic Ciprofloxacin given on Day 4, unless required sooner.
  Follow up visits occur on Days 5, 14 and 32.
  Interventions: Biological: Neisseria lactamica
- Group 2 (Experimental): Nasal drops containing Neisseria lactamica are administered at Day 0 by the study doctor.
  Follow up visits on Day 4 and 7 to check for N. lactamica carriage. Eradication therapy with the antibiotic Ciprofloxacin given on Day 14, unless required sooner.
  Follow up visits occur on Days 15, 24 and 42.
  Interventions: Biological: Neisseria lactamica

INTERVENTIONS:
Biological: Neisseria lactamica — Colonisation by bacteria is an immunising event; we proved this in humans by inoculating university students intranasally with the harmless commensal N. lactamica and we observed both specific systemic and mucosal antibody responses by 4 weeks. Experimental challenge with defined bacteria could tease out the Th17-mediated response mechanisms, which include waning of immunity over time, the induction of an incorrectly polarised T cell response, lack of cross-reactivity between strains or active immune evasion mechanisms employed by bacteria to subvert host immune effector mechanisms.

SUMMARY:
This study is part of a project that aims to develop a vaccine with N. lactamica that prevents meningitis. The investigators have previously given nose drops containing N. lactamica to over 340 volunteers, and shown that many of the volunteers (35-60%) become colonised without causing any illness or disease. In the future the investigators would like to modify N. lactamica so that it can carry vaccine molecules into the nose of children. To do this the investigators need to know more about the immune response generated against N. lactamica. Previously the investigators have shown that inoculation resulted in an immune (antibody) response in volunteers who were colonised. Taking an antibiotic called ciprofloxacin will treat N.lactamica in the nose and throat of the volunteers. The investigators need to know if the immune response to N. lactamica is the same when colonised volunteers are treated with the antibiotic after 4 days, is the same if the investigators treat volunteers after 14 days of carriage. This information will inform future studies.

DETAILED DESCRIPTION:
N. lactamica (Nlac) has been shown to be safe to use in human challenge experiments. Even at a very low dose of 10,000 colony forming units (cfu) long lasting colonisation with Nlac is easily induced in 35-65% of volunteers. The investigators have previously showed that increasing the inoculum to 100,000 cfu increased the subsequent carriage of Nlac to 50%. In 80-90% of those volunteers successfully colonised, this is detectable by 1-2 weeks.

Data regarding earlier detection of colonisation is currently lacking.

Colonisation has a clear effect on the volunteers nasal mucosal microbiome, in that meningococcal acquisition is effectively inhibited in volunteers who carry the organism. Colonisation is immunogenic, with an increase in specific serum IgG by 2 weeks and specific salivary IgA by 4 weeks.

No antibiotic eradication therapy has previously been given following experimental inoculation but Ciprofloxacin has been shown to be effective in the eradication of N. meningitidis.

To design future planned studies using Nlac nasal inoculation and colonisation in order to prevent invasive N. meningitidis disease, it is necessary to further evaluate the colonisation kinetics and efficacy of the eradication following antibiotic treatment. In previous challenges the investigators inoculated volunteers with Nlac and followed those volunteers for prolonged periods of time (over 6 months).

This study will compare the effect of short (4 days) versus longer (14 days) periods of nasal carriage of Nlac in volunteers on immunogenicity, and confirm the efficacy of antibiotic eradication therapy with ciprofloxacin.

Healthy adult volunteers will receive a nasal inoculation of Nlac with an antibiotic given on day 4 or 14. This information will be used to inform the design of future research into the colonisation and immunogenicity of related organisms.

Before designing future protocols the study investigators need to know whether a short containment of the volunteers will be sufficient for immunogenicity, and how quickly the volunteers can be discharged after antibiotic treatment.

A wild-type strain of Nlac (Y92-100) will be used for this study, selected because the investigators have previously used it safely in experimental challenge of over 340 human volunteers.

The same strain will be the parent strain for any future GMO work.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment
* Fully conversant in the English language
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Written informed consent to participate in the trial
* Willingness to take an antibiotic regimen after inoculation according to the study protocol
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and inoculation

Exclusion Criteria:

* Current active smokers
* N. lactamica or N. meningitidis detected on throat swab or nasal wash taken before the challenge
* Individuals who have a current infection at the time of inoculation
* Individuals who have been involved in other clinical trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period
* Individuals who have previously been involved in clinical trials investigating meningococcal vaccines or experimental challenge with N. lactamica
* Use of systemic antibiotics within the period 30 days prior to the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the inoculum
* Contraindications to the use of ciprofloxacin, specifically a history of epilepsy, prolonged QT interval, hypersensitivity to quinolones or a history of tendon disorders related to quinolone use
* Any clinically significant abnormal finding on clinical examination
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, for example recent surgery to the nasopharynx
* Occupational, household or intimate contact with immunosuppressed persons
* Pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Read, Principal Investigator — University of Southampton
Locations (1):
- Southampton NIHR Clinical Research Facility, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Evans CM, Pratt CB, Matheson M, Vaughan TE, Findlow J, Borrow R, Gorringe AR, Read RC. Nasopharyngeal colonization by Neisseria lactamica and induction of protective immunity against Neisseria meningitidis. Clin Infect Dis. 2011 Jan 1;52(1):70-7. doi: 10.1093/cid/ciq065. PMID 21148522
- [Derived] Dale AP, Theodosiou AA, Gbesemete DF, Guy JM, Jones EF, Hill AR, Ibrahim MM, de Graaf H, Ahmed M, Faust SN, Gorringe AR, Polak ME, Laver JR, Read RC. Effect of colonisation with Neisseria lactamica on cross-reactive anti-meningococcal B-cell responses: a randomised, controlled, human infection trial. Lancet Microbe. 2022 Dec;3(12):e931-e943. doi: 10.1016/S2666-5247(22)00283-X. PMID 36462524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers were recruited according to a REC approved recruitment strategy between 3/3/17 and 14/4/20. Participants attended a face to face screening visit at NIHR Southampton CRF to obtain informed consent and determine eligiblity
Pre-assignment Details: All enrolled participants were allocated to a group upon enrolment
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 13 | 8
Completed | 12 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Median (Full Range); unit: Years] | 33 [25 to 45] | 29 [25 to 39] | 31 [25 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 0 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Specific IgG titres [Median (Inter-Quartile Range); unit: Antibody titre] — Titres of specific antibodies in serum at baseline Population: Serological assessment only conducted in those participants in each group who were colonised and with serum samples available at each timepoint
  Antibody titre
    Nlac-specific IgG titre: number analyzed (Participants) | 6 | 6 | 12
    Nlac-specific IgG titre | 5.3 [3.3 to 6.4] | 4.6 [3.2 to 9.5] | 5.0 [3.0 to 7.5]
    Nmen-specific IgG titre: number analyzed (Participants) | 6 | 6 | 12
    Nmen-specific IgG titre | 22.6 [20.4 to 26.1] | 10.4 [8.0 to 13.9] | 17.1 [10.8 to 23.8]

OUTCOME MEASURES:

1. Primary Outcome: Measure the Antibodies, by Serological Antibody Titration, of Short Term Colonisation and Longer Colonisation
Description: Measure any rise in serological specific antibodies from samples taken at the start of the study (Day 0) and samples taken on Day 14 post inoculation and Day 28 post antibiotic eradication (Group 1 = Day 32 or Group 2 = Day 42)
Time Frame: Up to 42 Days
Population: Participants analysed are only those colonised in each group.
Measure: Median (Inter-Quartile Range); unit: Titres of antigen specific IgG
Groups:
- Day 0: Antigen specific IgG titres in serum prior to inoculation
- Day 14: Antigen specific IgG titres in serum 14 days after inoculation
- Eradication + 28: Antigen specific IgG titres in serum 28 days after eradication
Arm/Group | Day 0 | Day 14 | Eradication + 28
Number analyzed (Participants) | 6 | 6 | 6
Titres of antigen specific IgG
  Nlac-IgG Group 1 | 5.3 [3.3 to 6.4] | 5.5 [3.9 to 6.6] | 5.6 [4.6 to 7.1]
  Nlac-IgG Group 2 | 4.6 [3.2 to 9.5] | 13.4 [9.3 to 14.7] | 10.3 [7.7 to 13.1]
  Nmen-IgG Group 1 | 22.6 [20.4 to 26.1] | 23.7 [18.5 to 27.8] | 23.2 [19.4 to 26.6]
  Nmen-IgG Group 2 | 10.4 [8.0 to 13.9] | 17.3 [9.5 to 33.6] | 14.5 [9.5 to 22.3]

2. Secondary Outcome: Measure the Colonisation of Neisseria Lactamica
Description: Measure if Neisseria lactamica is able to colonise at or before Day 4 (for group 1) or Day 14 (for group 2) from cultured throat swabs.
Time Frame: Up to 14 Days
Population: Only those participants with at least one throat swab available at a post-challenge visit were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 13 | 7
Participants | 7 | 6

3. Secondary Outcome: Measure the Eradication of Neisseria Lactamica
Description: Record how successful eradication is up to Day 42, using throat swab samples.
Time Frame: Up to 42 Days
Population: Only includes those participants who were colonised at the visit at which they received antibiotic eradication
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 6 | 4
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: From enrolment until the end of follow up - 32 days post inoculation for Group 1 and 42 days post inoculation for Group 2
Description: Adverse events were reported for all enrolled participants for the duration of their involvement in the study and were defined as per the ClinicalTrials.gov definitions
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 3/13 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=13) | Group 2 (N=8)
Respiratory tract symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Malaise / lethargy / headache (General disorders) | 0 | 2 (3)
Diarrhoea / vomiting (Gastrointestinal disorders) | 0 | 1
Dysuria / cystitis (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT03549325/Prot_SAP_000.pdf